CLINICAL TRIAL: NCT04698083
Title: Retrospective Evaluation of Electrocardiographic Findings of Right Ventricular Overload in Covid 19 Patients With Respiratory Distress
Brief Title: Electrocardiographic QRS Axis Shift ,Rotation and COVİD-19
Status: Completed | Type: Observational
Sponsor: Ankara Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Şahbender Koç, Cardıologist, Ankara Education and Research Hospital
Other Study IDs: 22/7/2020-2152
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Group1:normal SpO2(NS,n = 80) and low SpO2(LS, n = 80).: Patients with normal oxygen saturation (SpO2; ≥ 90%) who did not receive oxygen therapy and patients with low SpO2(<90%) who received nasal oxygen therapy were included in this study
  Interventions: Diagnostic Test: Electrocardiography ,Tomographic imaging
- Group2:Rightward axis shift(Rws) and Leftward axis shift (Lws): Both groups were divided into two main subgroups:patients with Rws and patients with leftward shift(Lws) of the QRS axis.The patient numbers were as follows: NS Rws (n=37),NS Lws(n=43),LS Rws (n=40),andLS Lws (n=40)
  Interventions: Diagnostic Test: Electrocardiography ,Tomographic imaging

INTERVENTIONS:
Diagnostic Test: Electrocardiography ,Tomographic imaging — Based on electrocardiographic follow-up analyses,the two main groups were compared in terms of rotation condition (i.e., Cwr, normal transition, or CCwr), electrocardiographic intervals, and laboratory findings In our study,CO-RADS5 was considered an advanced tomographic finding(e.g., multifocal ground glass opacities with consolidation, vascular thickening,crazy paving pattern,mixed pattern),while CO-RADS1,2,3, and 4 were considered non-advanced tomographic findings.

SUMMARY:
In patients with coronavirus disease (COVID-19), severe dyspnea is the most dramatic complication.Severe respiratory difficulties may include electrocardiographic frontal QRS axis rightward shift (Rws) and clockwise rotation (Cwr).

This study investigated the predictability of advanced lung tomography findings with QRS axis shift and rotation.

This was a retrospective analysis of 160 patients.The patients were divided into two groups: normal oxygen saturation(SpO2) (NS; n = 80) and low SpO2(LS;n = 80).They were then divided into NS Rws (n = 37), NS leftward shift (Lws; n = 43), LS Rws (n = 40), and LS Lws (n = 40) according to electrocardiographic follow-up findings. These groups were compared in terms of electrocardiographic rotation (Cwr, counterclockwise rotation, or normal transition), tomographic stage (CO-RADS5(advanced)/CO-RADS1-4), electrocardiographic intervals, and laboratory findings

DETAILED DESCRIPTION:
The lung is the most seriously damaged organ in patients with coronavirus disease (COVID-19). In patients with advanced lung involvement, the alveoli are filled with fluid, white blood cells, mucus, and damaged lung cell debris [1].

The electrical position of the heart in the frontal plane is defined as normal, right, left, or northwest quadrant axis deviation, while its position in the horizontal plane is defined as clockwise rotation (Cwr), normal transition, or counterclockwise rotation (Ccwr)[2].

As respiratory disease progresses,rightward shift(Rws) of the frontal QRS axis can result from Cwr of the heart around its longitudinal axis as viewed from the apex, sudden increase in pulmonary vascular resistance causing right ventricle dilatation, or both [3].

Electrocardiographic changes should be monitored intermittently, as this disease progresses rapidly to near 50% mortality within 7-28 days [4].The aim of this study was to investigate whether easily detectable electrocardiographic axis and rotation changes could predict advanced lung involvement[4].

Methods Study design Records of 250 hospitalized patients with dyspnea and COVID-19 were analyzed retrospectively.Patients were excluded if they received positive pressurized oxygen therapy(n:25),underwent mechanical ventilation,(n:15)exhibited atrial fibrillation(n:10), conditions precluding the assessment of QRS transitional rotation ;complete bundle branch block(n:10), significant arrhythmias(n:5,complete atrioventricular block(n:2), polymorphic ventricular tachycardia(n:2), and ventricular fibrillation), Wolff-Parkinson-White syndrome(n:1), supraventricular tachycardia(n:4), or had unclear QRS axis orientation(n:20). The remaining160 patients who had electronic medical records, nursing records,at least three electrocardiographic recordings taken a few days apart, and laboratory and tomographic findings were included in the study.Patients with normal oxygen saturation (SpO2; ≥ 90%) who did not receive oxygen therapy and patients with low SpO2(<90%) who received nasal oxygen therapy were included in this study. Patients were divided into two groups: normal SpO2(NS,n = 80) and low SpO2(LS, n = 80).

Electrocardiographic measurements were performed as previously described.The Tpe (T peak to T end) interval was measured from precordial leads [5].The delta corrected QT interval(QTc) calculated as last electrocardiographic QTc minus first electrocardiographic QTc. Discrepancies between computerized electrocardiographic analysis and the mean of three computer-aided measurements(Adobe Photoshop program-300dpi resolution) by a researcher were resolved by consultation with a second researcher.

Using follow-up electrocardiography,according to the direction of QRS axis shift between the first and last electrocardiograms, both groups were divided into two main subgroups:patients with rightward shift (Rws) and patients with leftward shift(Lws) of the QRS axis.The patient numbers were as follows: NS Rws (n=37),NS Lws(n=43),LS Rws (n=40),andLS Lws (n=40). Based on electrocardiographic follow-up analyses,the two main groups were compared in terms of rotation condition (i.e., Cwr, normal transition, or CCwr), electrocardiographic intervals, and laboratory findings

Tomographic findings were evaluated in accordance with COVID-19 Reporting and Data System (CO-RADS)classification.CO-RADS scores are as follows: 1 (very low level of suspicion), 2 (low level of suspicion), 3 (equivocal), 4 (high level of suspicion),and 5 (very high level of suspicion)[6].

ELIGIBILITY:
Inclusion Criteria:

Hospitalized patients with dyspnea and COVID-19

Exclusion Criteria:

Patients who received positive pressurized oxygen therapy Patients who underwent mechanical ventilation, Atrial fibrillation Complete bundle branch block Significant arrhythmias(complete atrioventricular block, polymorphic ventricular tachycardia, and ventricular fibrillation), Wolff-Parkinson-White syndrome, supraventricular tachycardia Unclear QRS axis orientation.

-

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Hospitalized patients with dyspnea and COVID-19
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2020-07-22 (Actual); Primary Completion 2020-10-15 (Actual); Study Completion 2020-11-05 (Actual)

PRIMARY OUTCOMES:
Differences in the electrocardiographic QRS axis shift(°), | 10-15 days
  Differences in the axis shift between the Rws and Lws groups in patients with NS /LS groups.
Differences in the electrocardiographic rotation | 10-15 days
  Differences in clockwise,counterclockwise,normal transition between the groups.
Differences in the CO-RADS5/CO-RADS1-4 ratio | 10-15 days
  Differences in the CO-RADS5/CO-RADS1-4 ratio between the groups.

CONTACTS AND LOCATIONS:
Overall Officials: Şahbender Koç, Principal Investigator — University of Health Sciences Ankara Keçiören Education Hospital
Locations (1):
- Şahbender Koç, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Koc S, Bozkaya VO, Yikilgan AB. Electrocardiographic QRS axis shift, rotation and COVID-19. Niger J Clin Pract. 2022 Apr;25(4):415-424. doi: 10.4103/njcp.njcp_9_21. PMID 35439899